CLINICAL TRIAL: NCT04207749
Title: Clinical Evaluation of a Daily Wear Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-C018
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Refractive Errors; Myopia; Hyperopia
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID015385 (Experimental): LID015385 contact lenses worn at least 5 days per week and 8 hours per day in a daily wear modality (that is, not worn while sleeping) for approximately 3 months. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: LID015385 contact lenses; Device: CLEAR CARE
- Biofinity (Active Comparator): Comfilcon A contact lenses worn at least 5 days per week and 8 hours per day in a daily wear modality (that is, not worn while sleeping) for approximately 3 months. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: Comfilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: LID015385 contact lenses — Investigational soft contact lenses
  Arms: LID015385
Device: Comfilcon A contact lenses — Commercially available soft contact lenses
  Other Names: BIOFINITY®
  Arms: Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based cleaning and disinfecting solution

SUMMARY:
The purpose of this clinical study is to assess the safety and performance of an investigational soft contact lens compared to a commercially available soft contact lens when worn in a daily wear modality with frequent replacement.

DETAILED DESCRIPTION:
Subjects will attend 4 office visits: Screening/Baseline/Dispense; Week 1 Follow-up; Month 1 Follow-up; and Month 3 Follow-up/Exit. The total expected duration of participation for each subject is approximately 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Understand and sign an IRB/IEC approved Informed Consent form.
* Willing and able to attend all scheduled study visits and wear the assigned study lenses as required per protocol.
* Successful wear of frequent replacement, spherical, daily wear soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Manifest cylinder ≤ 0.75 diopter (D) in each eye.
* Best spectacle corrected visual acuity 20/20 or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Monovision contact lens wear.
* Any habitual wear of Biofinity lenses.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (18):
- United States (18):
  - Alcon Investigator 8103, Glendale, Arizona
  - Alcon Investigator 8101, Brentwood, California
  - Alcon Investigator 8102, Irvine, California
  - Alcon Investigator 8135, Los Angeles, California
  - Alcon Investigator 8108, Novato, California
  - Alcon Investigator 8062, Oakland, California
  - Alcon Investigator 8109, San Francisco, California
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6355, Orlando, Florida
  - Alcon Investigator 8115, Norcross, Georgia
  - Alcon Investigator 6567, Pittsburg, Kansas
  - Alcon Investigator 8063, Brighton, Massachusetts
  - Alcon Investigator 8100, New York, New York
  - Alcon Investigator 4817, Cleveland, Ohio
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 6401, Warwick, Rhode Island
  - Alcon Investigator 6353, Memphis, Tennessee
  - Alcon Investigator 8114, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 investigative sites located in the United States.
Pre-assignment Details: Of the 249 participants enrolled in this study, 15 were exited from the study as screen failures prior to randomization. This reporting group includes all randomized subjects/eyes (234/468).
Units Other Than Participants: eyes
Groups:
- Biofinity: Comfilcon A contact lenses worn at least 5 days per week and 8 hours per day in a daily wear modality (that is, not worn while sleeping) for approximately 3 months. CLEAR CARE was used for nightly cleaning and disinfection.
- LID015385: LID015385 contact lenses worn at least 5 days per week and 8 hours per day in a daily wear modality (that is, not worn while sleeping) for approximately 3 months. CLEAR CARE was used for nightly cleaning and disinfection.
Period: Overall Study
Arm/Group | Biofinity | LID015385
Started | 78; 156 eyes | 156; 312 eyes
Completed | 74; 148 eyes | 149; 298 eyes
Not Completed | 4; 8 eyes | 7; 14 eyes
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Unable to attend study visits due to COVID-19 pandemic | 1 | 4

BASELINE CHARACTERISTICS:
Population: Per Protocol (PP): All randomized subjects exposed to any study lenses evaluated in this study with at least one post-baseline (post-Dispense) contact lens corrected distance visual acuity (CLCDVA) assessment, minus all data/subjects that met any of the pre-defined critical deviation or evaluability criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofinity | LID015385 | Total
Number analyzed (Participants) | 75 | 145 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (8.2) | 31.3 (9.1) | 31.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 105 | 157
  Male | 23 | 40 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 72 | 139 | 211
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 65 | 95
  Black or African American | 2 | 1 | 3
  Chinese | 32 | 64 | 96
  Japanese | 6 | 7 | 13
  Korean | 4 | 7 | 11
  Other Asian | 0 | 1 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 75 | 145 | 220

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Contact Lens Corrected Distance Visual Acuity (CLCDVA) in Each Eye (CLL949-C018 + CLL949-C009)
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity.
Time Frame: Week 1 Follow-Up
Population: PP. A predefined subset of data from another similar completed study, CLL949-C009 (NCT03920280), was combined with this study to attain adequate power for the planned hypothesis testing of the primary and secondary outcome measures. The subset of subjects from CLL949-C009 that contributed data were those with Best-Corrected Visual Acuity (BCVA) of 20/20 or better in each eye at the Screening/Baseline/Dispense Visit.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 106 | 200
Number analyzed (eyes) | 212 | 400
logMAR | -0.06 (0.00) | -0.05 (0.00)
Statistical Analysis 1: Comparison: Biofinity vs LID015385; Test type: Non-Inferiority — Noninferiority in CLCDVA was declared if the upper confidence limit was less than 0.10 logMAR; Mixed effects repeated measures — Since noninferiority hypotheses are being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = 0.01, 95% CI 2-sided [-0.00 to 0.02] — Least squares mean difference (LID015385 minus Biofinity)

2. Secondary Outcome: Percentage of Subjects Achieving CLCDVA 20/20 or Better in Each Eye (CLL949-C018 + CLL949-C009)
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen, with 20/20 Snellen visual acuity considered normal distance eyesight.
Time Frame: Week 1 Follow-Up, at least 4 hours after lens insertion
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 106 | 200
percentage of subjects | 98.1 | 97.0
Statistical Analysis 1: Comparison: Biofinity vs LID015385; Test type: Non-Inferiority — Proportion of subjects is presented. Noninferiority in proportion of subjects achieving CLCDVA 20/20 or better in each eye was declared if the lower confidence limit was greater than -0.10; Farrington-Manning — [p-value comment as in outcome 1, analysis 1]; Difference in proportion = -0.01, 95% CI 2-sided [-0.06 to 0.04] — Lens difference (LID015385 minus Biofinity)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 3 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes were categorized under the actual study lenses exposed in the corresponding lens sequence.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- Biofinity - Ocular; Biofinity - Nonocular: Events reported in this group occurred while exposed to comfilcon A contact lenses
- LID015385 - Ocular; LID015385 - Nonocular: Events reported in this group occurred while exposed to LID015385 contact lenses
Arm/Group | Pretreatment | Biofinity - Ocular | Biofinity - Nonocular | LID015385 - Ocular | LID015385 - Nonocular
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/156 | 0/78 | 0/312 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/234 | 0/156 | 0/78 | 0/312 | 0/156
Other Adverse Events (participants affected / at risk) | 0/234 | 0/156 | 0/78 | 0/312 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT04207749/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT04207749/SAP_001.pdf